CLINICAL TRIAL: NCT03783650
Title: BP-CATCH: Boosting Primary Care Awareness and Treatment of Childhood Hypertension
Brief Title: Boosting Primary Care Awareness and Treatment of Childhood Hypertension
Acronym: BP-CATCH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely and will not resume due to the COVID-19 pandemic.
Sponsor: Montefiore Medical Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Rinke, Associate Professor of Pediatrics, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-9287; R01HS026239 (AHRQ)
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Pediatric Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): 0-6 months: Quality Improvement Collaborative (QIC) with PCP and without subspecialist, Registry & BP measurement 7-12 months: QIC with Subspecialist to improve communication and standardize, 13-18 months: Hub and Spoke co-management QIC with Primary care and Subspecialist 19-24 months: Sustainability of changes
  Interventions: Behavioral: QIC with PCP and without subspecialist; Behavioral: QIC with Subspecialist; Behavioral: Hub and Spoke co-management; Behavioral: Sustainability of changes
- Cohort 2 (Active Comparator): 0-6 months: Control condition Usual Care and Registry & BP measurement, 7-12 months: Quality Improvement Collaborative (QIC) with PCP and without subspecialist 13-18 months: QIC with Subspecialist to improve communication and standardize 19-24 months: Hub and Spoke co-management QIC with Primary care and Subspecialist
  Interventions: Behavioral: Control condition; Behavioral: QIC with PCP and without subspecialist; Behavioral: QIC with Subspecialist; Behavioral: Hub and Spoke co-management

INTERVENTIONS:
Behavioral: Control condition — Practices will submit control data and not receive centralized data feedback. They will also begin tracking data on a HTN registry and learn how to ensure accurate BP measurement is completed in their clinic.
  Arms: Cohort 2
Behavioral: QIC with PCP and without subspecialist — During this phase, practice will begin working on improving HTN practices within their clinic via a QIC, while the other cohort will act as a control (usual care) with data collection. They will attend an initial 1-day interactive video webinar learning session where they will learn QI methodology, enhance and practice QI skills, identify local 30-60 day aims to improve local HTN practices and increase their understanding of pediatric HTN. They will also begin tracking data on a HTN registry and learn how to ensure accurate BP measurement is completed in their clinic. They will participate in QI coaching, monthly video conferences, and monthly mini-root cause analyses (Mini-RCAs).
Behavioral: QIC with Subspecialist — Practices will integrate their HTN subspecialist into the QIC and focus on issues at the boundary of PCP and subspecialty care (e.g. pre-referral work-up, communication across providers, and time for next available appointment).
Behavioral: Hub and Spoke co-management — Practices will continue QIC components and implement a hub and spoke model, where the PCP diagnoses and provides definitive management for pediatric HTN with subspecialist support.
Behavioral: Sustainability of changes — Practices will sustain their changes, illustrating the durability of these system changes even after QIC completion and without central feedback and regular meetings.
  Arms: Cohort 1

SUMMARY:
The proposed research, building on an ongoing AHRQ-funded research project to prevent pediatric diagnostic errors in primary care (R01HS023608) and using a prospective, cluster-randomized, stepped wedge design, will investigate whether 1) a quality improvement collaborative (QIC) intervention without subspecialist involvement, 2) a QIC with subspecialists and primary care physicians (PCPs) mutually engaged, and/or 3) a hub and spoke co-diagnosis, co-management model where PCPs diagnose and manage pediatric hypertension (HTN) with a supporting subspecialist advisor, reduce errors in pediatric HTN diagnosis and management compared to each other and usual care.

DETAILED DESCRIPTION:
Pediatric HTN causes appreciable morbidity in pediatric patients and errors in diagnosis and management are frequent and understudied, jeopardizing pediatric safety in ambulatory settings. Additionally, the gap between the number of pediatric subspecialist providers and the number needed for patient care continues to widen, and it is unclear how to best reduce burden on subspecialists, improve PCP and subspecialist communication, and improve patient outcomes. This research team, with significant experience researching ambulatory pediatric safety, conducting QICs and HTN interventions, identified six large pediatric practice groups in rural, suburban and urban locations that are committed to reducing preventable HTN patient harm, to testing the effectiveness of a QIC to improve PCP HTN diagnosis and management, and to a hub and spoke HTN co-diagnosis and co-management model. The effect demonstrated by this project using a rigorous research design and the new 2017 pediatric HTN guidelines, will motivate pediatric clinics across the country to adopt these newly-identified best practices to improve pediatric HTN care. Primary care pediatricians have an imperative to diagnose and manage HTN and elevated BP (EBP) more accurately and earlier, and to improve interactions with subspecialists to reduce the lifelong preventable harm that results from these chronic conditions. This proposal, will identify a clear implementation strategy for rigorous, evidenced-based pediatric HTN diagnosis and management, and highlight a model to increase primary and subspecialty care integration that can be reproduced across other chronic conditions.

The primary human subjects of this work are the physicians and staff within the primary care pediatric practices and their associated pediatric hypertension subspecialists whose behavior the QIC is attempting to change. In order to know if these practices and subspecialists have changed their behaviors, we will look at patient data. To be included in the data cohort, patients must have a blood pressure (BP) measurement that is elevated (>= 90th percentile for patient's sex, age, and height, or >=120/80 (regardless of sex/age/ height) at a healthcare maintenance visit or non-acute care visit (e.g. chronic disease follow-up visit). The following patients would be excluded from the data cohort:

* Prior hypertension or elevated BP diagnosis. Patient can have prior elevated BP measurements as long as no diagnosis has been made
* BP>95th percentile + 30mm or >180/120 or symptomatic patient
* Prior diagnosis of congenital heart disease, chronic kidney disease, urologic disease (e.g. posterior urethral valve, vesicoureteral reflux) or organ transplant,
* Previously included in BP-CATCH data entry
* Acute care visit (e.g., fever, viral illness, asthma attack, pain in any body part, etc.)

ELIGIBILITY:
Inclusion:

* Primary care pediatric practices who see children ages 3-22 years old.
* Practice must be able to field a 3-person core improvement team who can participate in the quality improvement collaborative.

Exclusion:

- Non-pediatric practices

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Number of patients without all correct diagnostic and management decisions | average 34 months
  Number of patients without all correct diagnostic and management decisions per 100 patients with measured elevated BP

SECONDARY OUTCOMES:
Number of patients without re-measuring of BP twice in clinic via auscultation | average 34 months
  Number of patients without re-measuring of BP twice in clinic via auscultation at specified points per 100 patients with measured elevated BP
Number of patients without weight counseling management decisions | average 34 months
  Number of patients without weight counseling at specified points per 100 patients with measured elevated BP
Number of patients without lifestyle modification counseling management decisions | average 34 months
  Number of patients without lifestyle modification counseling management decisions at specified points per 100 patients with measured elevated BP
Number of patients without nutrition counseling management decisions | average 34 months
  Number of patients without nutrition counseling management decisions at specified points per 100 patients with measured elevated BP
Number of patients without repeat BP measurement visits appropriately timed | average 34 months
  Number of patients without repeat BP measurement visits appropriately timed at specified points per 100 patients with measured elevated BP
Number of patients without initial laboratory workup diagnostic decisions | average 34 months
  Number of patients without initial laboratory workup at specified points per 100 patients with measured elevated BP
Number of patients without Subspecialist referral | average 34 months
  Number of patients without Subspecialist referral at specified points per 100 patients with measured elevated BP
Number of patients without echocardiogram workup diagnostic decisions | average 34 months
  Number of patients without echocardiogram workup diagnostic decisions at specified points per 100 patients with measured elevated BP
Number of patients without echocardiogram diagnostic decisions | average 34 months
  Number of patients without echocardiogram diagnostic decisions at specified points per 100 patients with measured elevated BP
Number of patients without radiology diagnostic decisions | average 34 months
  Number of patients without radiology diagnostic decisions at specified points per 100 patients with measured elevated BP
BPs measured correctly that met specific criteria | average 34 months
  Number of measured BPs correctly per 100 patients with BP measured with appropriately screened patient, patient position, cuff size, inflation, BP percentiles correctly documented and interpreted
Time to third new next available subspecialist appointment | average 33 months
  Third new next available appointment for pediatric patients to subspecialist clinics in order to assess the effects of pediatric primary care providers referring and managing different types of patients with hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Rinke, MD, Principal Investigator — Albert Einstein College of Medicine and The Children's Hospital at Montefiore
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heo M, Rea CJ, Brady TM, Bundy DG, Melikam ES, Orringer K, Tarini BA, Giuliano K, Twombley K, Goilav B, Kelly P, Faith MS, Pietrobelli A, Rinke ML. Racial and Ethnic Disparities in Pediatric Counseling on Nutrition, Lifestyle, and Weight: A Secondary Analysis of the BP-CATCH Randomized Clinical Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2456238. doi: 10.1001/jamanetworkopen.2024.56238. PMID 39878982
- [Derived] Rea CJ, Brady TM, Bundy DG, Heo M, Faro E, Giuliano K, Goilav B, Kelly P, Orringer K, Tarini BA, Twombley K, Rinke ML. Pediatrician Adherence to Guidelines for Diagnosis and Management of High Blood Pressure. J Pediatr. 2022 Mar;242:12-17.e1. doi: 10.1016/j.jpeds.2021.11.008. Epub 2021 Nov 10. PMID 34774574